CLINICAL TRIAL: NCT02888717
Title: Concordance Study of Molecular Biology Analysis for Para-aortic Nodes in the Ultra-staging of Advanced Cervical Cancers (GYNOSNA)
Brief Title: Molecular Biology Analysis for Para-aortic Nodes in the Ultra-staging of Advanced Cervical Cancers
Acronym: GYNOSNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-N-2014-06
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Advanced Cervical Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OSNA stadification during surgery (Experimental): The para-aortic dissection surgery is performed in the usual way. The lymph nodes are isolated from fat tissue during surgery, and will be analysis both by histological analysis and OSNA analysis
  Interventions: Procedure: 'OSNA stadification during surgery'

INTERVENTIONS:
Procedure: 'OSNA stadification during surgery' — The para-aortic dissection surgery is performed in the usual way. The lymph nodes are isolated from fat tissue during surgery, and cut into 4 slices sterile.
  * Slices A and C are sent OSNA analysis
  * Slices B and D are sent ultimately histological analysis (1 cup HES or 5 cup HES + IHC) The nodes of less than 5 mm will be sent in final histological analysis due to the inability to cut into 4.
  After the analysis, the report indicates whether the node is:
  * Free (-): <250 copies
  * Micrometastatic (+): 250 ≤ - <5,000 copies,
  * Macrometastatic (++): ≥ 5000 copies.

SUMMARY:
The para-aortic lymph node involvement in the advanced stage of cervical cancer is a poor prognostic factor for overall survival. Concomitant chemo-radiotherapy has become the standard treatment for advanced cervical cancer. In case of para-aortic lymph node involvement, an extension of radiotherapy fields is recommended.

A prospective multicentre study shown that the survival rate of patients with node ≤ 5 mm and which benefited from the expansion of radiotherapy fields was identical to the survival of pN0 patients.

However, due to a specific disease, this technique should not be performed in all patients. It is necessary to reliably select patients with retroperitoneal lymph node involvement. For this, it is recommended that prior to the concurrent chemo-radiotherapy, nodal staging surgery with a definitive histological analysis.

So we propose to use molecular diagnostic test OSNA (One Step Nucleic Acid Amplification) to improve lymph node metastasis detection sensitivity to achieve ultra-staging compared to conventional histology.

DETAILED DESCRIPTION:
The para-aortic lymph node involvement in the advanced stage of cervical cancer is a poor prognostic factor for overall survival. Concomitant chemoradiotherapy has become the standard treatment for advanced cervical cancer. In case of para-aortic lymph node involvement, an extension of radiotherapy fields is recommended.

A prospective multicenter study shown that the survival rate of patients with node ≤ 5 mm and which benefited from the expansion of radiotherapy fields was identical to the survival of pN0 patients.

However, due to a specific disease, this technique should not be performed in all patients. It is necessary to reliably select patients with retroperitoneal lymph node involvement. For this, it is recommended that prior to the concurrent chemoradiotherapy, nodal staging surgery with a definitive histological analysis.

So we suggest using molecular diagnostic test OSNA (One Step Nucleic Acid Amplification) to improve lymph node metastasis detection sensitivity to achieve ultra-staging compared to conventional histology.

We propose to consider a new concordance study to assess the feasibility of the technical OSNA in a new indication: cervical cancer.

The analysis protocol of a concordance study is the same regardless of the location of the cancer. We evaluate the use of OSNA in order to ultrastaging of lymph node involvement for patients with advanced cancer of the cervix.

Our hypothesis is that OSNA would be:

* better than the usual histological staging method
* and equivalence in terms of sensitivity and specificity compared to intensive histological method To complete this study we propose to search the initial brain tumor expression of cytokeratin 19.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 or over
2. Cervical cancer of any histological type
3. Cervical cancer of advanced stage (>= IB2)
4. negative para-aortic routine PET CT scan
5. Patient affiliated to a social protection scheme
6. Information on the study delivered to the patient

Exclusion Criteria:

1. Patients minor
2. Patient pregnant or breastfeeding or of childbearing age without effective contraception
3. Other concurrent cancer or history of cancer (in the 5 years preceding the entry into the trial), except in situ cervical cancer treated basal cell or squamous cell or treated carcinoma
4. Legal incapacity or limited legal capacity. medical or psychological conditions not allowing the subject to understand the study and sign the consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
compare the performance of OSNA for the detection of lymph node metastases in advanced cervical cancer | 15 days between surgery and OSNA results
  The main objective is to compare the performance of OSNA to both conventional methods and intensive histological analysis, for the detection of lymph node metastases in advanced cervical cancer.
  The evaluation criteria is :
  * Determination of number of lymph node metastases expressed in a size in mm for conventional and intensive histological analysis.
  * Determination of the number of lymph node metastases expressed in a number of copies in molecular biology.

CONTACTS AND LOCATIONS:
Overall Officials: JAFFRE Isabelle, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- ICO René Gauducheau, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No